CLINICAL TRIAL: NCT05533450
Title: A Multicenter Randomized Controlled Study on the Efficacy and Safety of Multi-focal Scleral Contact Lens in the Treatment of Ultra-high Myopia in Children and Adolescents
Brief Title: A Study on the Efficacy and Safety of Multi-focal Scleral Contact Lens
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shandong University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: kjb-gmj-v1.1-20220814
Record Dates: First submitted 2022-09-05; First posted 2022-09-09 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: High Myopia
Keywords: high myopia; children and adolescents; defocus; scleral contact lens

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-focal rigid scleral contact lens (Experimental): During the study period, subjects will wear a multi-focal rigid scleral contact lens daily.
  Interventions: Device: Multi-focal rigid scleral contact lens
- Rigid gas permeable contact lens (Active Comparator): During the study period, the subjects will wear rigid contact lenses daily
  Interventions: Device: Rigid gas permeable contact lens

INTERVENTIONS:
Device: Multi-focal rigid scleral contact lens — True scleral lenses rest on the sclera and do not touch the cornea and limbus, leaving a clear area between the contact lens and the cornea.
  Other Names: OVCTEK
  Arms: Multi-focal rigid scleral contact lens
Device: Rigid gas permeable contact lens — RGP contact lens is designed from a special rigid hydrophobic material. Patients wear RGP contact lens to form a "contact lens-tear-cornea" system to correct irregular astigmatism, reduce aberrations, provide good visual quality, and control the development of the disease through mild "shaping" effect.
  Other Names: OVCTEK
  Arms: Rigid gas permeable contact lens

SUMMARY:
The rigid scleral contact lens with optical multi-focal design adopted in this study can focus the light in part of the optical area on the front of the retina to form myopic defocus, in order to delay the axial changes in children and adolescents with ultra-high myopia. In this study, RGP was used as a control, and a multicenter, randomized, controlled trial was conducted to verify the safety and effectiveness of multifocal scleral contact lenses for the correction of ultra-high myopia in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to understand and sign the informed consent when accompanied by parents or guardians.
2. Age from 8 years old to15 years old.
3. The equivalent spherical lens of both eyes after ciliary muscle paralysis is -5.00D to -20.00D, the astigmatism is ≤-3.50D.
4. Willing to wear hard contact lenses, and able to wear only the hard contact lenses provided by the study as required and ensure adequate wearing duration.

(6) Best corrected visual acuity of both eyes ≥ 0.8.

Exclusion Criteria:

(1) Allergic or intolerant to rigid contact lens or its care products or ciliary muscle paralysis drugs.

Strabismus and/or amblyopia. (3) Those who have worn hard contact lenses in the past 30 days are using atropine, defocus frame lens, bifocal lens or progressive lens, acupuncture, etc. for myopia treatment.

(4) Any clinically significant active eye disease, such as glaucoma, uveitis, chorioretinitis, central retinal artery or vein occlusion, and so on.

(5) Patients with systemic diseases that may affect the wearing of hard contact lenses, such as hyperthyroidism, diabetes, mental illness, and so on.

(6) are using drugs that affect their eye health. (7) History of eye injury or surgery. (8) Incapacitated or unable to follow the visitor as required. (9) Other conditions not suitable for inclusion as judged by the investigator.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2022-10-18 (Estimated); Primary Completion 2022-10-18 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Axial length | 2 years
  Two-year change in axial length

SECONDARY OUTCOMES:
changes of spherical equivalent | 2 years
  Spherical equivalent as measured by cycloplegia autorefraction

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Eye Disease Prevention & Treatment Center, Shanghai, Shanghai Municipality
  - Shanghai Eye Disease Prevention and Treatment Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No